CLINICAL TRIAL: NCT04419649
Title: A Phase 2, Open-Label, Ascending Dose Study of KER-050 for the Treatment of Anemia in Patients With Very Low, Low, or Intermediate Risk Myelodysplastic Syndromes (MDS)
Brief Title: A Study of Elritercept to Treat Anemia in Adults With Very Low, Low, or Intermediate Risk Myelodysplastic Syndromes (MDS)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KER050-MD-201; 2023-507469-24-00 (EU CTIS Number)
Record Dates: First submitted 2020-06-03; First posted 2020-06-05 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Myelodysplastic Syndromes; Cytopenia
Keywords: Transfusion; Drug Therapy; Elritercept; TAK-226; KER-050
MeSH Terms: conditions — Myelodysplastic Syndromes; Cytopenia

STUDY DESIGN:
Intervention Model Description: Ascending dose study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Part 1: Elritercept Cohort 1 (Experimental): Participants will be administered elritercept at 0.75 milligrams per kilogram (mg/kg), subcutaneous (SC) injection, every 4 weeks on Day 1 of each cycle for up to 4 cycles (each cycle = 28 days). Following the above dose regimen, participants will continue to receive elritercept, administered SC, on Day 1, every 4 weeks up to 24 cycles (each cycle = 28 days).
  Interventions: Drug: Elritercept
- Part 1: Elritercept Cohort 2 (Experimental): Participants will be administered elritercept at 1.5 mg/kg, SC injection, every 4 weeks on Day 1 of each cycle for up to 4 cycles (each cycle = 28 days). Following the above dose regimen, participants will continue to receive elritercept, administered SC, on Day 1, every 4 weeks up to 24 cycles (each cycle = 28 days).
  Interventions: Drug: Elritercept
- Part 1: Elritercept Cohort 3 (Experimental): Participants will be administered elritercept at 2.5 mg/kg, SC injection, every 4 weeks on Day 1 of each cycle for up to 4 cycles (each cycle = 28 days). Following the above dose regimen, participants will continue to receive elritercept, administered SC, on Day 1, every 4 weeks up to 24 cycles (each cycle = 28 days).
  Interventions: Drug: Elritercept
- Part 1: Elritercept Cohort 4 (Experimental): Participants will be administered elritercept at 3.75 mg/kg, SC injection, every 4 weeks on Day 1 of each cycle for up to 4 cycles (each cycle = 28 days). Following the above dose regimen, participants will continue to receive elritercept, administered SC, on Day 1, every 4 weeks up to 24 cycles (each cycle = 28 days).
  Interventions: Drug: Elritercept
- Part 1: Elritercept Cohort 5 (Experimental): Participants will be administered elritercept at 5.0 mg/kg, SC injection, every 4 weeks on Day 1 of each cycle for up to 4 cycles (each cycle = 28 days). Following the above dose regimen, participants will continue to receive elritercept, administered SC, on Day 1, every 4 weeks up to 24 cycles(each cycle = 28 days).
  Interventions: Drug: Elritercept
- Part 2: Elritercept Dose Confirmation Cohort A (Experimental): Participants with ring sideroblasts (RS)-positive Myelodysplastic syndrome (MDS) who are requiring red blood cell (RBC) transfusions will be administered Elritercept at 3.75 mg/kg, SC injection, on Day 1, every 4 weeks for up to 24 cycles (each cycle = 28 days). The dose can be modified based on participant's response.
  Interventions: Drug: Elritercept
- Part 2: Elritercept Dose Confirmation Cohort B (Experimental): Participants with non-RS MDS who are requiring RBC transfusions will be administered Elritercept at 3.75 mg/kg, SC injection, on Day 1, every 4 weeks for up to 24 cycles (each cycle = 28 days). The dose can be modified based on participant's response.
  Interventions: Drug: Elritercept
- Part 2: Elritercept Dose Confirmation Cohort C (Experimental): Participants who are non-transfused with either RS-positive MDS or non-RS MDS will be administered Elritercept at 3.75 mg/kg, SC injection, on Day 1, every 4 weeks for up to 24 cycles (each cycle = 28 days). The dose can be modified based on participant's response.
  Interventions: Drug: Elritercept
- Experimental: Part 2: Elritercept Dose Confirmation Cohort D (Experimental): Participants with chronic myelomonocytic leukemia (CMML) and anemia will be administered Elritercept at 3.75 mg/kg, SC injection, on Day 1, every 4 weeks for up to 24 cycles (each cycle = 28 days). The dose can be modified based on participant's response.
  Interventions: Drug: Elritercept
- Part 2: Elritercept Dose Confirmation Cohort E (Experimental): Participants with MDS (either RS-positive or non-RS) who are requiring RBC transfusions, have iron-overload, and are receiving iron chelation therapy will be administered Elritercept at 3.75 mg/kg, SC injection, on Day 1, every 4 weeks for up to 24 cycles (each cycle = 28 days). The dose can be modified based on participant's response.
  Interventions: Drug: Elritercept
- Part 2: Elritercept Dose Confirmation Cohort F (Experimental): Participants with MDS (either RS-positive or non-RS) who are requiring RBC transfusions, have iron-overload, and are not receiving iron chelation therapy will be administered Elritercept at 3.75 mg/kg, SC injection, on Day 1, every 4 weeks for up to 24 cycles (each cycle = 28 days). The dose can be modified based on participant's response.
  Interventions: Drug: Elritercept
- Part 2: Elritercept Dose Confirmation Cohort G (Experimental): Participants with MDS (either RS-positive or non-RS) who require RBC transfusions and have either relapsed, become refractory to, or intolerant to frontline luspatercept treatment will be administered Elritercept at 3.75 mg/kg, SC injection, on Day 1, every 4 weeks for up to 24 cycles (each cycle = 28 days). The dose can be modified based on participant's response.
  Interventions: Drug: Elritercept
- Long-term Extension Cohort (Experimental): Participants from Part 1 and 2 cohorts who may have potential benefit from continued elritercept treatment, in the opinion of the Investigator, may elect to continue in the LTE at the same dose they were being administered in Part 1 and 2, SC injection, on day 1, every 4 weeks until end of treatment (EOT) (approximately 122 months).
  Interventions: Drug: Elritercept

INTERVENTIONS:
Drug: Elritercept — Elritercept SC injection.
  Other Names: KER-050; TAK-226

SUMMARY:
The main aim of this study is to learn how safe elritercept is and how well adults with anemia associated with lower-risk MDS tolerate treatment with different doses of elritercept. Other aims are to learn how safe elritercept is by looking at how many participants have MDS that worsens during the study and learn about the effects of elritercept on anemia linked to MDS. The study will also look to learn how elritercept affects the production of healthy RBCs.

DETAILED DESCRIPTION:
Elritercept (KER-050) is a recombinant fusion protein being studied to increase red blood cell production by inhibiting the signaling of a subset of the transforming growth factor beta (TGF-ß) family of proteins.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information in accordance with national and local study participant privacy regulations.
2. Male or female ≥ 18 years of age, at the time of signing informed consent.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 (if related to anemia).
4. Females of childbearing potential and sexually active males must agree to use highly effective methods of contraception.
5. In the opinion of the Investigator, the participant is able and willing to comply with the requirements of the protocol (e.g., all study procedures, return for follow-up visits).

Part 1 Inclusion Criteria

Participants are eligible to be included in Part 1 of the study only if all the following criteria apply:

1. Diagnosis of MDS according to WHO classification that meets International Prognostic Scoring System-Revised (IPSS-R) classification of very low, low, or intermediate risk disease.
2. Less than (<)5percent (%) blasts in bone marrow during the Pretreatment Period.
3. Peripheral blood white blood cell (WBC) count <13,000/microliter (μL) during the Pretreatment Period.
4. Anemia defined as:

   1. In non-transfused participants, having received no RBC transfusions within 8 weeks, Hgb concentration ≤ 10.0 g/dL during the Pretreatment Period OR
   2. In LTB participants, having received 1 to 3 units of RBCs for Hgb ≤ 9.0 g/dL within 8 weeks of the Pretreatment Period.

      OR
   3. In HTB participants, having received ≥ 4 units of RBCs for Hgb ≤ 9.0 g/dL within 8 weeks of the Pretreatment Period.

Part 1 Extension - Abbreviated Inclusion Criteria

Participants from Part 1 are eligible to be included in Part 1 Extension of the study only if all the following criteria apply:

1. Previously completed 4 cycles of elritercept in Part 1 with no dose-limiting toxicities (DLTs).
2. Participant has the potential to benefit from administration of elritercept, in the opinion of the Investigator.
3. < 5% blasts in bone marrow.
4. Peripheral WBC count < 13,000/μL during the 28 days prior to cycle 5 day 1 (C5D1).

Part 2 Inclusion Criteria

Participants are eligible to be included in Part 2 of the study only if all the following criteria apply:

1. Cohort A:

   * Diagnosis of MDS according to WHO classification that meets IPSS-R classification of very low, low, or intermediate risk disease.
   * ring sideroblast (RS)-positive as defined by WHO 2016 criteria.
   * Requiring at least 2 units of RBC transfusions in the preceding 8 weeks before cycle 1 day 1 (C1D1).
2. Cohort B:

   * Diagnosis of MDS according to WHO classification that meets IPSS-R classification of very low, low, or intermediate risk disease.
   * Non-RS as defined by WHO 2016 criteria.
   * Requiring at least 2 units of RBC transfusions in the 8 weeks before C1D1.
3. Cohort C:

   * Diagnosis of MDS according to WHO classification that meets IPSS-R classification of very low, low, or intermediate risk disease.
   * Has anemia, defined by Hgb ≤ 10 g/dL during the Pretreatment Period, and received no RBC transfusion in the 8 weeks before C1D1.
4. Cohort D:

   * Diagnosis of CMML according to WHO classification.
   * Has anemia, defined by Hgb ≤ 10 g/dL during the Pretreatment Period, and received no RBC transfusion in the 8 weeks before C1D1.
   * OR
   * Received at least 2 units of RBC transfusions for anemia in the 8 weeks before C1D1.
5. Cohort E:

   * Diagnosis of MDS according to WHO classification that meets IPSS-R classification of very low, low, or intermediate risk disease.
   * Requiring ≥ 2 units of RBC transfusions in the preceding 8 weeks before C1D1.
   * Receipt of ≥ 20 units of RBC in transfusion over the participant's lifetime.
   * Serum ferritin > 1000 nanograms per milliliter (ng/mL) on ≥ 2 assessments in the preceding 8 weeks before C1D1.
   * Treated with stable dose of iron chelation therapy for ≥ 8 weeks prior to C1D1.
6. Cohort F:

   * Diagnosis of MDS according to WHO classification that meets IPSS-R classification of very low, low, or intermediate risk disease.
   * Requiring ≥ 2 units of RBC transfusions in the preceding 8 weeks before C1D1.
   * Receipt of ≥ 20 units of RBC in transfusion over the participant's lifetime.
   * Serum ferritin > 1000 ng/mL on ≥ 2 assessments in the preceding 8 weeks before C1D1.
   * Not treated with iron chelation therapy in the preceding 8 weeks before C1D1 and not eligible to initiate iron chelation therapy in the opinion of the Investigator and in accordance with local treatment guidelines for initiation of iron chelation therapy.
7. Cohort G:

   * Diagnosis of MDS according to WHO classification that meets IPSS-R classification of very low, low, or intermediate risk disease.
   * RS-positive as defined by WHO 2016 criteria OR non-RS as defined by WHO 2016 criteria.
   * Relapsed, refractory, or intolerant to frontline luspatercept treatment and have not received an interceding therapy (for example, erythropoiesis-stimulating agent [ESA])

     * Relapsed is defined as documentation of response to luspatercept therapy and subsequent development of a need for transfusion(s).
     * Refractory is defined as documentation of no response with luspatercept ≥ 1 mg/kg administered for ≥ 12 weeks duration.
     * Intolerant is defined as documentation of discontinuation of luspatercept therapy due to intolerance or an AE at any time after introduction.
   * Requiring ≥ 2 units of RBC transfusions over 8 weeks prior to C1D1.
   * Erythropoietin (EPO) < 500 international units per liter (U/L) at Baseline.
   * Last dose of luspatercept is ≥ 3 weeks and < 12 months from C1D1.
8. < 5% blasts in bone marrow assessed by bone marrow aspirate during the Pretreatment Period.

Part 1 Exclusion Criteria

Participants are excluded from Part 1 of the study if any of the following criteria apply.

Medical History

1. Diagnosis of MDS with deletion of chromosome 5q (Del5q).
2. Active infection requiring parenteral antibiotic therapy within 28 days prior to C1D1 or oral antibiotics within 14 days of C1D1. Prophylactic antibiotics and/or antifungals for neutropenia are allowed.
3. Presence of uncontrolled heart disease or New York Heart Association (NYHA) Class III or IV heart failure.
4. History of drug or alcohol abuse (as defined by the Investigator) within the past 2 years.
5. History of stroke, deep venous thrombosis (DVT), or arterial embolism within 6 months prior to C1D1.
6. Major surgery within 28 days prior to C1D1. Participants must be completely recovered from any previous surgery prior to C1D1.
7. Known positive for human immunodeficiency virus (HIV), active infectious hepatitis B virus (HBV), or active infectious hepatitis C virus (HCV). Participants without known positive history of HIV, HBV, and/or HCV do not require further testing, unless testing is mandated per local guidelines.
8. Any malignancy other than MDS that has not been in remission and/or has required systemic therapy including radiation, chemotherapy, hormonal therapy, or surgery, within 1 year prior to C1D1. Diagnosis of secondary MDS (i.e., MDS known to have arisen as the result of chemical injury or treatment with chemotherapy and/or radiation for other diseases).
9. History of solid organ or hematological transplantation.
10. Presence of uncontrolled hypertension, defined as systolic blood pressure (BP) ≥ 150 mmHg or diastolic BP ≥ 100 mmHg despite adequate treatment.
11. Body mass index (BMI) ≥ 40 kilograms per meter square (kg/m^2) during the Pretreatment Period.
12. History of severe allergic or anaphylactic reaction(s) or hypersensitivity to recombinant proteins or excipients in the investigational medicinal product (IMP).

Treatment History

1. Prior treatment with azacitidine, decitabine, lenalidomide, luspatercept, or sotatercept.
2. Treatment with ESA within 56 days prior to C1D1.
3. Prior or concurrent chronic treatment with granulocyte colony-stimulating factor (G-CSF) or granulocyte-macrophage colony-stimulating factor (GM-CSF).
4. Iron chelation therapy if initiated within 8 weeks prior to C1D1.
5. Vitamin B12 therapy initiated within 8 weeks prior to C1D1. Participants on stable replacement doses for ≥ 8 weeks and without concurrent vitamin B12 or folate deficiency are allowed.
6. Treatment with another investigational drug or device or approved therapy for investigational use ≤ 28 days prior to C1D1, or, if the half-life of the previous product is known, within 5 times the half-life prior to C1D1, whichever is longer.

Laboratory Exclusions (during Pretreatment Period)

1. Platelet count > 450 ✕ 10^9/L or < 30 ✕ 10^9/L.
2. Transferrin saturation < 15%.
3. Ferritin < 50 nanograms per milliliter (ng/mL).
4. Folate < 4.5 nanomoles per liter (nmol/L) (< 2.0 ng/mL).
5. Vitamin B12 < 148 picomoles per liter (pmol/L) (< 200 picograms per milliliter [pg/mL]).
6. Estimated glomerular filtration rate (GFR) < 30 milliliter per minute per 1.73 meter square (mL/min/1.73 m^2), as determined by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.
7. Positive for HIV.

Miscellaneous

1. Pregnant or lactating females.
2. Any other condition not specifically noted above which, in the opinion of the Investigator, would preclude the participant from participating in the study.
3. Participants who are investigational site staff members directly involved in the conduct of the trial and their immediate family members, site staff members otherwise supervised by the Investigator, or participants who are Sponsor or contract research organization (CRO) employees directly involved in the conduct of the study. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.

Part 1 Extension - Exclusion Criteria

Participants from Part 1 are excluded from Part 1 Extension of the study if any of the following criteria apply.

Medical History

1. Discontinuation of IMP in Part 1 for any reason.
2. Has not completed a study visit in the past 12 months.
3. Active infection requiring parenteral antibiotic therapy within 28 days prior to C5D1 or oral antibiotics within 14 days of C5D1. Prophylactic antibiotics and/or antifungals for neutropenia are allowed.
4. Presence of uncontrolled heart disease or NYHA Class III or IV heart failure.
5. History of drug or alcohol abuse (as defined by the Investigator) within the past 2 years.
6. History of stroke, DVT, or arterial embolism within 6 months prior to C5D1.
7. Major surgery within 28 days prior to C5D1. Participants must be completely recovered from any previous surgery prior to C5D1.
8. Known positive for HIV, active infectious HBV, or active infectious HCV. Participants without known positive history of HIV, HBV, and/or HCV do not require further testing, unless testing is mandated per local guidelines.
9. Any malignancy other than MDS that has not been in remission and/or has required systemic therapy including radiation, chemotherapy, hormonal therapy, or surgery, within 1 year prior to C5D1.
10. History of solid organ or hematological transplantation.
11. Presence of uncontrolled hypertension, defined as systolic BP ≥ 150 mmHg or diastolic BP ≥ 100 mmHg despite adequate treatment.
12. BMI ≥ 40 kg/m^2 during the 28 days prior to C5D1.

Treatment History

1. Prior treatment with azacitidine, decitabine, lenalidomide, luspatercept, or sotatercept.
2. Treatment with ESA within 56 days prior to C5D1.
3. Prior or concurrent chronic treatment with G-CSF or GM-CSF.
4. Iron chelation therapy if initiated within 8 weeks prior to C5D1.
5. Vitamin B12 with treatment initiated within 8 weeks prior to C5D1. Participants on stable replacement doses for ≥ 8 weeks and without concurrent vitamin B12 or folate deficiency are allowed.
6. Treatment with another investigational drug or device or approved therapy for investigational use ≤ 28 days prior to C5D1, or, if the half-life of the previous product is known, within 5 times the half-life prior to C5D1, whichever is longer. Previous treatment with elritercept is acceptable.

Laboratory Exclusions (during Abbreviated Pretreatment Period)

1. Platelet count > 450 × 10^9/L or < 30 × 10^9/L.
2. Transferrin saturation < 15%.
3. Ferritin < 50 ng/mL.
4. Folate < 4.5 nmol/L (< 2.0 ng/mL).
5. Vitamin B12 < 148 pmol/L (< 200 pg/mL).
6. Estimated GFR < 30 mL/min/1.73 m^2, as determined by the CKD-EPI equation.

Miscellaneous

1. Pregnant or lactating females.
2. Any other condition not specifically noted above which, in the opinion of the Investigator, would preclude the participant from participating in the study.
3. Participants who are investigational site staff members directly involved in the conduct of the trial and their immediate family members, site staff members otherwise supervised by the Investigator, or participants who are Sponsor or CRO employees directly involved in the conduct of the study. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.

Part 2 Exclusion Criteria

Participants are excluded from Part 2 of the study if any of the following criteria apply.

Medical History

1. Diagnosis of MDS with Del5q.
2. Diagnosis of secondary MDS (i.e., MDS known to have arisen as the result of chemical injury or treatment with chemotherapy and/or radiation for other diseases).
3. Active infection requiring parenteral antibiotic therapy within 28 days prior to C1D1 or oral antibiotics within 14 days of C1D1. Prophylactic antibiotics and/or antifungals for neutropenia are allowed.
4. Presence of the following cardiac conditions:

   1. Presence of uncontrolled heart disease or NYHA Class III or IV heart failure.
   2. QTcF (QT interval corrected by Fridericia's formula) > 500 msec on the screening or C1D1 electrocardiogram (ECG; mean of 3 measurements).
   3. Uncontrolled clinically significant arrhythmia (participants with rate-controlled atrial fibrillation are not excluded).
   4. Acute myocardial infarction or unstable angina pectoris ≤ 6 months prior to C1D1.
5. Presence of uncontrolled hypertension, defined as systolic BP ≥ 160 mmHg or diastolic BP ≥ 100 mmHg despite adequate treatment.
6. History of stroke, DVT, or arterial embolism within 6 months prior to C1D1.
7. History of drug or alcohol abuse (as defined by the Investigator) within the past 2 years.
8. Major surgery within 28 days prior to C1D1. Participants must be completely recovered from any previous surgery prior to C1D1.
9. Any malignancy other than MDS or CMML that has not been in remission and/or has required major surgery or systemic therapy including radiation, chemotherapy, targeted therapy, or hormonal therapy within 1 year prior to C1D1.
10. History of solid organ or hematological transplantation.
11. Diagnosis of hemolytic anemia, active bleeding, hemoglobinopathies, or congenital disorders as a cause of the participant's anemia.
12. NCI-CTCAE Grade ≥ 2 bleeding events within the 3 months prior to C1D1.
13. Receipt of an RBC or platelet transfusion for any reason(s) or combination of reasons other than underlying MDS within the 16 weeks prior to C1D1. If a participant requires a transfusion for an unanticipated reason during the Pretreatment Period, a prolonged screening period may be considered after discussion with the Medical Monitor.
14. Known positive for HIV, active infectious HBV with positive viral load (HBV DNA), or active infectious HCV with positive viral load (HCV RNA). Participants without known positive history of HIV, HBV, and/or HCV do not require further testing, unless testing is mandated per local guidelines.
15. BMI ≥ 40 kg/m^2.
16. History of severe allergic or anaphylactic reaction(s) or hypersensitivity to recombinant proteins or excipients in the IMP.
17. Diagnosis of cirrhosis, non-alcoholic steatohepatitis, alcoholic liver disease, hepatitis, or other liver disease (acute or chronic) meeting Child-Pugh C criteria for hepatic impairment. Participants with elevated liver enzymes are allowed if the liver enzyme elevation is suspected to be due to iron-overload or iron chelation, and other hepatic causes have been ruled out, in the opinion of the Investigator.

Treatment History

1. Prior treatment with azacitidine, decitabine, lenalidomide, or sotatercept.
2. Prior treatment with luspatercept (Cohorts A, B, C, D, E, and F only).
3. Treatment with ESA within 8 weeks prior to C1D1.
4. Prior or concurrent chronic treatment with G-CSF or GM-CSF, for reasons other than for treatment of MDS.

   a. Note: Previous treatment with G-CSF or GM-CSF for MDS, which has been discontinued ≥ 8 weeks prior to C1D1 is allowed.
5. Iron chelation therapy if initiated within 8 weeks prior to C1D1. Participants on stable doses of iron chelation therapy for ≥ 8 weeks are allowed.
6. Vitamin B12 and/or folate therapy initiated within 8 weeks prior to C1D1. Participants on stable replacement doses for ≥ 8 weeks and without concurrent vitamin B12 or folate deficiency are allowed.
7. Any need to receive a prohibited medication.
8. Treatment with another investigational drug or device or approved therapy for investigational use within 8 weeks prior to C1D1, or, if the half-life of the previous product is known, within 5 times the half-life prior to C1D1, whichever is longer.

Laboratory Exclusions (during Pretreatment Period)

1. Peripheral WBC count ≥ 13,000/μL.
2. Platelet count > 450 × 10^9/L or < 25 × 10^9/L.
3. Transferrin saturation < 15%.
4. Ferritin < 50 ng/mL.
5. Folate < 4.5 nmol/L (< 2.0 ng/mL).
6. Vitamin B12 < 148 pmol/L (< 200 pg/mL).
7. Estimated GFR < 30 mL/min/1.73 m^2 as determined by the CKD-EPI equation.

Miscellaneous

1. Pregnant or lactating females.
2. Any other condition not specifically noted above which, in the opinion of the Investigator, would preclude the participant from participating in the study.
3. Participants who are investigational site staff members directly involved in the conduct of the trial and their immediate family members, site staff members otherwise supervised by the Investigator, or participants who are Sponsor or CRO employees directly involved in the conduct of the study. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.

For Cohort G ONLY:

1. Any luspatercept related AE Grade ≥ 3 that has not resolved to baseline or Grade ≤ 1.
2. No history of allergy/anaphylaxis/hypersensitivity to luspatercept.
3. No prior treatment with imetelstat.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-08-19 (Actual); Primary Completion 2029-10-30 (Estimated); Study Completion 2031-10-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | From treatment initiation to end of study (up to 11.2 years)
  An AE is defined as any untoward medical occurrence, in a clinical study participant administered a medicinal product, that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not it is related to the medicinal (investigational) product. An SAE is any untoward medical occurrence that, at any dose: results in death, is life threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a medically important event.

SECONDARY OUTCOMES:
Number of Participants with Progression to Higher Risk MDS or Acute Myeloid Leukemia (AML) | From study day 1 through end of study (up to 11.2 years)
  The progression to higher risk MDS or AML will be assessed as per the World Health Organization (WHO) 2016 criteria.
Percentage of Participants with Low Transfusion Burden (LTB) and High Transfusion Burden (HTB) who Achieve RBC Transfusion Independence (TI) | From study day 1 through end of study (up to 11.2 years)
  Participants with LTB and HTB achieving RBC TI greater than or equal to (≥) 8 weeks, overall RBC TI and based on RS status will be assessed.
Percentage of Participants who Achieve Hematologic Improvement Erythroid (HI-E) Response Based on Modified 2006 International Working Group (IWG) | From study day 1 to end of study (up to 11.2 years)
  The response is defined as a mean hemoglobin (Hgb) increase of ≥1.5 grams per deciliter (g/dL) from Baseline during any 8-week period during the treatment period for LTB participants and participants with non-transfused anemia, and is defined as a reduction by ≥ 4 units of RBCs transfused during any 8-week period on study compared with the 8-week period prior to study cycle 1 day 1 (C1D1) (cycle length = 28 days) for HTB participants. Participants achieving overall HI-E response and based on RS status will be assessed.
Percentage of Participants who Achieve Overall Erythroid Response | Up to approximately 11.2 years
  The response is defined as a mean hemoglobin (Hgb) increase of ≥1.5 grams per deciliter (g/dL) from Baseline during any 8-week period during the treatment period for LTB participants and participants with non-transfused anemia, and is defined as a reduction by ≥ 4 units of RBCs transfused during any 8-week period on study compared with the 8-week period prior to study cycle 1 day 1 (C1D1) (cycle length = 28 days) for HTB participants. TI is defined as RBC transfusion independence for ≥ 8 weeks. Overall erythroid response is defined as HI-E or TI over any 8-week period. Participants achieving overall erythroid response and based on RS status will be assessed.
Percentage of Participants who Achieve Erythropoietic Improvement | Up to approximately 11.2 years
  The improvement is defined as a mean Hgb increase of ≥1.5 g/dL from Baseline for ≥14 days (in the absence of RBC transfusions) for LTB participants and participants with non-transfused anemia and is defined as a reduction of ≥50% or ≥4 RBC units transfused compared with pretreatment over an 8-week period for HTB participants. Participants achieving overall improvement and based on RS status will be assessed.
Mean Change from Baseline in Hgb | Baseline, multiple timepoints post treatment up to 11.2 years
  At each visit, the mean of the change from baseline in Hgb will be calculated across participants.
Time to HI-E Response | Up to approximately 11.2 years
  The response is defined as a mean hemoglobin (Hgb) increase of ≥1.5 grams per deciliter (g/dL) from Baseline during any 8-week period during the treatment period for LTB participants and participants with non-transfused anemia, and is defined as a reduction by ≥ 4 units of RBCs transfused during any 8-week period on study compared with the 8-week period prior to study cycle 1 day 1 (C1D1) (cycle length = 28 days) for HTB participants.
Duration of HI-E Response | Up to approximately 11.2 years
  The response is defined as a mean hemoglobin (Hgb) increase of ≥1.5 grams per deciliter (g/dL) from Baseline during any 8-week period during the treatment period for LTB participants and participants with non-transfused anemia, and is defined as a reduction by ≥ 4 units of RBCs transfused during any 8-week period on study compared with the 8-week period prior to study cycle 1 day 1 (C1D1) (cycle length = 28 days) for HTB participants.
Time to TI Response | Up to approximately 11.2 years
  TI is defined as RBC transfusion independence for ≥ 8 weeks.
Duration of TI response | Up to approximately 11.2 years
  TI is defined as RBC transfusion independence for ≥ 8 weeks.
Percentage of LTB and HTB Participants who Achieve TI | Weeks 12, 16, 24 and 48
Number of Participants with Change from Baseline in Red Cell Parameters | Up to approximately 11.2 years
  The red cell parameters including reticulocyte count, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), and reticulocyte cell Hgb will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (47):
- United States (5):
  - City of Hope National Medical Center, Duarte, California
  - University of Miami School of Medicine Sylvester Comprehensive Cancer Center (SCCC), Miami, Florida
  - H. Lee Moffitt Cancer Center and Research Center, Tampa, Florida
  - Karmanos Cancer Institute at Mclaren Greater Lansing, Lansing, Michigan
  - University of Pittsburgh Medical Health Center, Pittsburgh, Pennsylvania
- Australia (12):
  - Border Medical Oncology Research, Albury, New South Wales
  - Tweed Hospital, Tweed Heads, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Townsville University Hospital, Douglas, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Boxhill Hospital, Box Hill, Victoria
  - University Hospital Geelong, Geelong, Victoria
  - Austin Health, Heidelberg, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - St Vincent's Hospital Melbourne, Melbourne, Victoria
  - Ballarat Oncology & Haematology Service, Wendouree, Victoria
- Czechia (3):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Vseobecna Fakultni Nemocnice Praha, Prague
- France (7):
  - CHU Angers - Hopital Hotel Dieu, Angers
  - Centre Hospitalier de la Region dAnnecy, Épagny
  - CHU de Nantes - Hotel Dieu, Nantes
  - CHU Nice - Hopital de l'Archet 1, Nice
  - Hopital Saint-Louis, Paris
  - CH Rene-Dubos, Pontoise
  - CHU de Bordeaux - Hopital Haut-Leveque, Talence
- Germany (11):
  - Klinikum Bayreuth GmbH, Bayreuth
  - Charite-Campus Benjamin Franklin, Berlin
  - Praxis am Volkspark Berlin, Berlin
  - University Hospital Bonn, Bonn
  - Marien Hospital Dusseldorf GMBH, Düsseldorf
  - Universitaetsklinikum Duesseldorf AoeR, Düsseldorf
  - Klinikum Esslingen GmbH, Esslingen am Neckar
  - University Hospital Halle (Saale), Halle
  - Universitaetsklinikum Leipzig AoeR, Leipzig
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz, Mainz
  - Universitaetsmedizin Rostock, Rostock
- Israel (2):
  - Sheba Medical Center - Sheba Fund for Health Services and Research, Ramat Gan
  - Sourasky Medical Center - Infrastructure and Health Services Fund of the Tel Aviv Medical Center, Tel Aviv
- Middlemore Hospital, Auckland, New Zealand
- Spain (6):
  - Hospital Universitario Central de Asturias, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - ICO l'Hospitalet - Hospital Duran i Reynals, Barcelona
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.